CLINICAL TRIAL: NCT06068933
Title: K-HEARS MCI: Hearing Health Care for Korean American Older Adults With Mild Cognitive Impairment - Pilot
Brief Title: Hearing Health for Korean American Older Adults With Mild Cognitive Impairment
Acronym: K-HEARS MCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is being terminated due to insufficient participant recruitment within the projected timeframe
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00249500; R56DC019686 (NIH)
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Age-related Hearing Impairment; Personal Communication; Mild Cognitive Impairment
MeSH Terms: conditions — Communication; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants in Phase 2-A MCI Focused Trial will be randomized into a two arms: immediate intervention and delayed intervention. Participants in Phase 2-B KA Older Adult Focused Trial will not be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 2A -MCI Pilot Trial Immediate Treatment Group (Experimental): Immediate treatment with K-HEARS intervention
  Interventions: Behavioral: K-HEARS Intervention; Device: K-HEARS Sound Amplifier Intervention
- Phase 2A -MCI Pilot Trial Delayed Treatment Group (Placebo Comparator): 6-month delayed treatment with K-HEARS intervention
  Interventions: Behavioral: K-HEARS Intervention; Device: K-HEARS Sound Amplifier Intervention
- Phase 2B -KA Older Adult Focused Trial (non-randomized) (Other): Immediate treatment with K-HEARS intervention
  Interventions: Behavioral: K-HEARS Intervention; Device: K-HEARS Sound Amplifier Intervention

INTERVENTIONS:
Behavioral: K-HEARS Intervention — Tailored aural rehabilitation for participant and care partner
Device: K-HEARS Sound Amplifier Intervention — Tailored fitting and programming of a personal sound amplifier. This will be accompanied by a component of aural rehabilitation.

SUMMARY:
The objective of this study is to develop and assess the feasibility, acceptability, and preliminary efficacy of a community-delivered, affordable, and accessible hearing care intervention tailored to the needs of community-dwelling Korean American (KA) older adults with mild cognitive impairment (MCI) and their care partners that integrates a low-cost over-the-counter amplification device and hearing rehabilitation through a randomized controlled pilot study. Each dyad will consist of the study participant and their care partner.

DETAILED DESCRIPTION:
The study consists of three phases: 1) Phase 1: development of the intervention through exploratory focus groups and/or semi-structured interviews and prototyping via open-labeled trial 2) Phase 2A: randomized, controlled pilot study with study participants randomized to an immediate treatment group, versus a 6-month delayed treatment group of an intervention specific for individuals with MCI, 3) Phase 2B: a non-randomized pragmatic-focused trial of community-dwelling older KAs with hearing loss but without MCI, and 4) Phase 3: qualitative evaluation of the experience and supplemental feedback through exploratory focus groups and/or semi-structured interviews.

ELIGIBILITY:
PARTICIPANT INCLUSION CRITERIA FOR PHASE 2A: MCI-Pilot Trial

* Age ≥ 60 years
* Self-identified as first-generation Korean American
* Self-reported ability to read and speak Korean
* Hearing loss identified by screening audiometry pure-tone-average (PTA) 1, 2, 4 kilohertz > 25 decibel hearing loss in better hearing ear
* Mild cognitive impairment (CDR=0.5 and/or Korean Montreal Cognitive Assessment (MoCA-K) <23)
* Report not currently using a hearing aid
* Has a care partner able to participate in the study
* Stable medication regimen. Stable (for 2 weeks or longer) dosing of medication (e.g. antidepressants, antipsychotics) for neuropsychiatric symptoms

PARTICIPANT INCLUSION CRITERIA FOR PHASE 2B: KA Older Adult-focused Trial:

* Age ≥ 60 years
* Self-identified as first-generation Korean American
* Self-reported ability to read and speak Korean
* Hearing loss identified by screening audiometry pure-tone-average (PTA) 1, 2, 4 kilohertz >= 35 decibel Hearing Loss in better hearing ear
* Report not currently using a hearing aid
* Has a care partner able to participate in the study

CARE PARTNER INCLUSION CRITERIA (same for both Phase 2A and 2B)

* Age 18 years or older
* Able to read and speak Korean
* Lives in the same household with the participant or has at least daily interactions
* Aural-oral verbal communication as primary communication modality
* Able to accompany participant to all study visits

EXCLUSION CRITERIA (same for both Phase 2A and 2B)

Participant exclusion criteria

* Residence in an assisted living facility (ALF) or nursing home (NH)
* Medical contraindication to use of amplification device (e.g., draining ear)
* Currently using a hearing aid or listening device

Care partner exclusion criteria

• Individuals who do not fulfill inclusion criteria

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE-S) score | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Score range 0-40. 0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap.

SECONDARY OUTCOMES:
Revised UCLA Loneliness Scale | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Score is the sum of 20-item self-reported measure. Scores range from 20 to 80.
  Score ranges:
  20-34 - Low degree of loneliness 35-49 - Moderate degree of loneliness 50-64 - Moderately high degree of loneliness 65-80 - High degree of loneliness.
Short Form-12 (SF-12) Mental Component Score | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  The 12-Item Short Form Survey (SF-12) measures the construct of self-reported health-related quality of life. Score ranges from 0-100 with higher scores indicating better mental health functioning.
Social Network size Measured by Lubben Social Network Index | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Measures social network size for both family and friends and also the frequency of interaction with them. Higher scores indicate higher level of social engagement. Score range (0-30).

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, RN, Principal Investigator — JHU School Of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States